CLINICAL TRIAL: NCT00735878
Title: A Phase I/II Pharmacokinetic and Pharmacodynamic Study of ABT-751 in Combination With Carboplatin in Patients With Advanced Lung Cancer
Brief Title: Pharmacokinetic & Pharmacodynamic Study of ABT-751 With Carboplatin in Patients With Advanced Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: data from a similar did not show efficacy.
Sponsor: Konstantin Dragnev (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor-Investigator, Konstantin Dragnev, Associate Professor Hematology/Oncology, Dept of Med, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0412
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer
Keywords: Lung Cancer; Advanced Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — ABT751; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ABT-751 100 mg and Carboplatin (Experimental): 100 mg BID ABT-751 orally for 7 days. Carboplatin AUC 4.5 once every 21 days.
  Interventions: Drug: ABT-751 and Carboplatin
- ABT-751 125 mg and Carboplatin (Experimental): 125 mg BID ABT-751orally for 7 days. Carboplatin AUC 4.5 or 6 once every 21 days.
  Interventions: Drug: ABT-751 and Carboplatin
- ABT-751 150 mg and Carboplatin (Experimental): 150 mg BID ABT-751orally for 7 days. Carboplatin AUC 6 once every 21 days.
  Interventions: Drug: ABT-751 and Carboplatin

INTERVENTIONS:
Drug: ABT-751 and Carboplatin — This primary objective of this Phase 1/2 study is to evaluate the DLT and MTD of escalating oral doses of ABT-751 given BID on Day 1 of each cycle for 7 days in combination with carboplatin given on a 21-day schedule. The carboplatin dose is fixed at AUC 6 and will be administered on Day 4 during the first cycle to facilitate the pharmacokinetic analysis. During the subsequent cycles both agents will be administered on Day 1. ABT-751 is administered at the following dose levels using the Simon rapid dose escalation model: 100, mg, 125 mg, 150 mg, 175 mg and 200 mg BID.
  Other Names: Paraplatin

SUMMARY:
Primary Objectives:

The primary objectives of this study are as follows:

• To determine the dose limiting toxicity (DLT) and the maximum tolerated dose (MTD) of escalating ABT-751 in combination with fixed dose carboplatin in patients with advanced non small cell lung cancer (NSCLC).

• To evaluate the efficacy of the combination with ABT-751 and carboplatin in patients with advanced NSCLC

• To determine the median survival in the study population

Secondary Objectives

The secondary objectives are:

• To characterize the pharmacokinetic profile of ABT-751 given in combination with carboplatin in a subset of patients, treated at the MTD or recommended doses for Phase 2.

• To determine the pharmacodynamics of ABT-751 as a single agent and the combination of ABT-751 and carboplatin as evaluated by cell cycle analysis of buccal mucosa cells.

DETAILED DESCRIPTION:
This primary objective of this Phase 1/2 study is to evaluate the DLT and MTD of escalating oral doses of ABT-751 given BID (twice daily) on Day 1 of each cycle for 7 days in combination with carboplatin given on a 21-day schedule. The carboplatin dose is fixed at AUC 6 and will be administered on Day 4 during the first cycle to facilitate the pharmacokinetic analysis. During the subsequent cycles both agents will be administered on Day 1. ABT-751 is administered at the following dose levels using the Simon rapid dose escalation model: 100, mg, 125 mg, 150 mg, 175 mg and 200 mg BID.

Initially, 1 patient will be enrolled in dose level 1. If the patient experiences a Grade 2 toxicity, an additional 2 patients will be enrolled at the same dose level. If 1 of the 3 patients experiences a Grade 3 (or higher toxicity), the cohort will be expanded to 6 patients. However, if 1 patient completes one cycle at the assigned dose regimen without experiencing a Grade 2 toxicity, enrollment in the next cohort (dose level 2) can begin. This rapid dose escalation scheme will apply to cohorts 1 through 3.

Initially, in the 4th cohort (dose level 4), a minimum of three patients will be enrolled. If 1 of the 3 patients experiences a Grade 3 (or higher toxicity), the cohort will be expanded to 6 patients. However, if 3 patients complete one cycle at the assigned dose regimen without experiencing a Grade 3 (or higher toxicity), enrollment in the next cohort (dose level 5) can begin. This scheme will apply to cohorts 4, 5, and 6 MTD is defined as the highest dose of ABT-751 given in combination with carboplatin at which fewer than 33% of patients experience DLT. MTD will be evaluated at the end of the first cycle (21 days). Toxicities will be determined also at the end of cycle 2 to evaluate the safety of combining both agents on day 1. If the MTD has not been determined after completion of the 6th cohort (dose level 6), based on an overall review of toxicity at each cohort, the Investigator may select a dose thought to be the recommended dose for Phase 2 studies. Six patients treated at MTD will undergo PK (pharmacokinetic) and PD (pharmacodynamic) evaluation. An additional cohort of 14-20 patients will be enrolled at either the MTD or at the recommended Phase 2 dose level administering both drugs on day 1. During this portion of the study patients will be withdrawn from the study if any of the following occur:

• Patient or patient's legally acceptable representative decides to withdraw consent.

• Patient's response to therapy is unsatisfactory, as evidenced by progression of disease as defined by RECIST Criteria for Tumor Response (within 2 cycles)

• The patient experiences toxicities deemed possibly or probably related to drug that have not resolved to at least Grade 2 or lower within three weeks.

• The patient requires more than one dose reduction because of toxicities attributable to ABT-751.

• The patient requires during the study period alternate antineoplastin agent, concurrent radiotherapy or surgery of the only measurable site(s) of disease.

• The patient becomes pregnant or begins to breast-feed.

• The investigator believes it is in the best interest of the patient to discontinue study drug administration.

If grade 3 or higher toxicities develop in 2 or more out of the first 6 patients who receive both drugs on day 1 on a dose level at which no such toxicities were noted on the ABT-751 day 1/carboplatin day 4 schedule, the additional patients for the second portion of the study will receive the latter schedule.

If toxicities characteristic of carboplatin (myelosuppression and others) are observed at the AUC 6 dose, carboplatin dose will be lowered to AUC 4.5 and the following dose escalation schema will be employed, beginning at the same ABT-751 dose as the one at which the toxicity developed:

All patients should receive antiemetics prior to carboplatin. A regimen of dexamethasone 10 mg and dolasetron 100 mg IV prior to carboplatin infusion may be used.

The study enrollment will be limited to patients with advanced NSCLC. Treatment will continue until progression of disease, unacceptable toxicities or withdrawal of informed consent. Male and female cancer patients will be selected to participate in the study according to the selection criteria.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Pathologically or cytologically confirmed diagnosis of NSCLC .
3. At least one measurable lesion (not amenable to resection) for Response Evaluation Criteria in Solid Tumors (RECIST) tumor assessments. Target lesions must not have been in the previous radiation port.
4. Advanced stage of disease (IIIB with malignant pleural effusion or Stage IV) with no known curative treatment that has progressed despite therapy for recurrent/metastatic disease or prior therapy was discontinued due to intolerable toxicities. During the phase II portion of the study, previously untreated patients with IIIB with malignant pleural effusion or Stage IV NSCLC may be enrolled.
5. For patients participating in the phase I part of the study, no alternative therapy is available that is expected to prolong overall or progression-free survival. Unacceptable toxicities during first- or second-line therapy or evidence for disease progression.
6. Adequate hematologic, renal and hepatic function as follows:

   * Hematologic: ANC (absolute neutrophil count) ≥ 1200/mm3; Platelets; ≥ 100,000/mm3; hemoglobin: ≥ 8.5 g/dL;
   * Renal function: serum creatinine ≤ 2.0 mg/dL; renal (CrCl > 50 ml/min by Jelliffe or Cockcroft Gault Formula),
   * Hepatic function: Bilirubin ≤ 2.0 mg/dL (≤ 3.0 mg/dL for patients with liver metastases); AST (aspartate aminotransferase) and ALT (alanine aminotransferase) ≤ 2.5 X the upper limits of normal (ULN) (≤ 5 X ULN for patients with liver metastases).
7. Adequate performance status, Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-1.
8. Prior platinum (cisplatin, carboplatin or oxaliplatin) therapy is allowed.
9. Patient or patient's legally acceptable representative has voluntarily signed and dated an informed consent form approved by an Institutional Review Board (IRB), prior to any study-specific procedures.

Exclusion Criteria:

1. Any other malignancy within 3 years except in situ carcinoma.
2. Untreated central nervous system (CNS) metastasis.
3. A greater than Grade 1 National Cancer Institute Common Toxicity Criteria (NCI CTC) neurology category findings at baseline.
4. Concurrent anti-cancer therapy or radiotherapy.
5. Concurrent therapy with colchicines.
6. Prior therapy with ABT-751.
7. Cytotoxic chemotherapy within 3 weeks of initiating investigational treatment.
8. Any investigational therapy within 4 weeks.
9. Female patients that are pregnant or breastfeeding.
10. Patients of childbearing potential (male and female) that do not agree to use a contraceptive method deemed acceptable by the investigator while in the study and for up to three months following completion of therapy.
11. Documented allergy or hypersensitivity to carboplatin or sulfa.
12. Patient has received more than 2 prior chemotherapy regimens for advanced disease. Adjuvant chemotherapy administered more than 6 months prior to enrollment does not count towards this limit.
13. Patient is classified as 3 or 4 by New York Heart Association (NYHA) Functional Classification, defined as:

    - Class 3: Patients with marked limitation of physical activity, comfortable at rest, but less than ordinary activity causes symptoms.

    - Class 4: Patients are unable to carry on any physical activity without symptoms and symptoms are present even at rest.
14. Evidence of clinically significant medical condition(s) that compromises safety, compliance, or study conduct, and/or is considered by the investigator to be unable to tolerate the proposed treatment or procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin H Dragnev, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Ma T, Fuld AD, Rigas JR, Hagey AE, Gordon GB, Dmitrovsky E, Dragnev KH. A phase I trial and in vitro studies combining ABT-751 with carboplatin in previously treated non-small cell lung cancer patients. Chemotherapy. 2012;58(4):321-9. doi: 10.1159/000343165. Epub 2012 Nov 12. PMID 23147218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants will be recruited from inpatient and outpatient populations at DHMC and through physician referrals.
Groups:
- 100 mg; 125 mg; 150 mg: Maximum Tolerated Dose Determination Phase
Period: Phase I- Dose Determination
Arm/Group | 100 mg | 125 mg | 150 mg
Started | 1 (13 subjects enrolled. One subject withdrew consent prior to receiving therapy & was replaced.) | 7 | 5
Completed | 1 (12 subjects received at least one cycle of treatment and were evaluable per the protocol.) | 7 | 4
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Phase II- Determined Dose
Arm/Group | 100 mg | 125 mg | 150 mg
Started | 0 | 7 | 0
Completed | 0 (Seven subjects completed therapy within the Phase II portion of the trial.) | 7 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 mg | 125 mg | 150 mg | Total
Number analyzed (Participants) | 1 | 14 | 5 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 9 | 3 | 13
  >=65 years | 0 | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 | 62 (7.65) | 63 (9.28) | 62 (8.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 4 | 7
  Male | 1 | 11 | 1 | 13
Region of Enrollment [Number; unit: participants]
  United States | 1 | 14 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of ABT-751 in Combination With Carboplatin
Description: The maximum tolerated dose (MTD) of escalating ABT-751 in combination with fixed dose Carboplatin AUC 6 in patients with advanced non small cell lung cancer (NSCLC). Initially, 1 patient will be enrolled in dose level 1. If the patient experiences a Gr 2 toxicity, additional 2 patients will be enrolled at the dose level. If 1 of the 3 patients experience a Gr 3 toxicity or higher the cohort will be expanded to 6 patients. However, if 1 patient completes one cycle at the assigned dose regimen without a Gr 2 toxicity, enrollment in the next cohort (dose level 2) can begin. The rapid dose escalation scheme will apply to cohorts 1 through 3.
Time Frame: 21 Days (end of cycle 1)
Measure: Number; unit: mg of ABT-751
Groups:
- Group 1/ Dose Escalating ABT-751 in Combination With Carboplat: Oral dose escalating of ABT-871 given BID on Day 1 of each cycle for 7 days in combination with Carboplatin given on a 21-day schedule. There will be up to 7 Cohorts(Dose Levels) from 100 to 200 mg/m2 of ABT-751 mg BID with Carboplatin AUC 4.5 for the first two cohorts, and AUC 6 for the remaining.
Arm/Group | Group 1/ Dose Escalating ABT-751 in Combination With Carboplat
Number analyzed (Participants) | 13
mg of ABT-751 | 125

2. Primary Outcome: Objective Response Rate of Participants Using A Combination of ABT-751 and Carboplatin
Description: The effectiveness of the combination with ABT-751 and carboplatin in patients with advanced NSCLC as measured by objective response rate. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) for target lesions and assessed by CT or MRI: Complete Response (CR), The disappearance of all known disease determined by two observations not less than four weeks apart.; Partial Response (PR), At least a 30% or more decrease in total tumor load of the lesions that have been measured to determine the effect of therapy by two observations not less than four weeks apart.; Overall Response (OR) = CR + PR
Time Frame: 42 days (end of cycle 2)
Measure: Count of Participants; unit: Participants
Groups:
- Group 1/ Dose Escalating ABT-751 in Combination With Carboplat: Oral dose escalating of ABT-871 given BID on Day 1 of each cycle for 7 days in combination with Carboplatin given on a 21-day schedule. There will be up to 7 Cohorts(Dose Levels) from 100 t0 200 mg/m2 of ABT-751 mg BID
Arm/Group | Group 1/ Dose Escalating ABT-751 in Combination With Carboplat
Number analyzed (Participants) | 13
Participants | 13

3. Primary Outcome: The Median Survival in the Study Population
Description: Median overall survival using the Kaplan Meier method
Time Frame: from the start of the study until the last subject dies (up to 100 weeks)
Population: 12 Participants were enrolled into the phase 1 portion of the tiral and later 8 more patients were enrolled for a total of 20 analyzed patients.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Participants Treated at MTD: Median overall survival of all patients (Ph I and Ph II) treated at MTD.
Arm/Group | All Participants Treated at MTD
Number analyzed (Participants) | 20
months | 11.7 [5.9 to 27.0]

4. Secondary Outcome: Pharmacokinetic Profile of ABT-751 for Phase 2
Description: The pharmacokinetic profile of ABT-751 given in combination with carboplatin in a subset of patients, treated at the MTD or recommended doses for Phase 2.
Time Frame: Randomization to maximum tolerated dose confirmed
Population: Data were not collected. The PK analysis was not performed at the request of financial sponsor.
Groups:
- Group 1/ Dose Escalating ABT-751 in Combination With Carboplat: Oral dose escalating of ABT-871 given BID on Day 1 of each cycle for 7 days in combination with Carboplatin given on a 21-day schedule. There will be up to 7 Cohorts(Dose Levels) from 100 to 200 mg/m2 of ABT-751 mg BID
- Group 2/ Phase II: Phase 2 participants treated at MTD.
Arm/Group | Group 1/ Dose Escalating ABT-751 in Combination With Carboplat | Group 2/ Phase II
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Patients With Buccal Cells Demonstrating a Decline in Cyclin D1
Description: Cyclin D1 levels were evaluated by immunoblot analyses of pretreatment (day 0) and paired posttreatment (day 4, 8 and 22) buccal swabs.
Time Frame: pretreatment (Day 0) and patient paired post- treatment (Days 4,8, 22) buccal swabs.
Population: A subset of patients treated at the recommended Phase II dose from Phase II/Group 2
Measure: Number; unit: participants
Groups:
- Phase II/Group 2: Number of participants evaluated for buccal mucosa cells
Arm/Group | Phase II/Group 2
Number analyzed (Participants) | 6
participants
  Decline in Cyclin D1 expression on Day 4 | 0
  Decline in Cyclin D1 expression on Day 8 | 3
  Decline in Cyclin D1 expression on Day 22 | 4

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | 100 mg | 125 mg | 150 mg
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/14 | 1/5
Other Adverse Events (participants affected / at risk) | 1/1 | 12/14 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg (N=1) | 125 mg (N=14) | 150 mg (N=5)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg (N=1) | 125 mg (N=14) | 150 mg (N=5)
Constipation (Gastrointestinal disorders) | 0 (0) | 5 (5) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 3 (3) | 3 (3)
Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes